CLINICAL TRIAL: NCT02847988
Title: Facilitating Functional Independence in Patients Receiving Prolonged Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RML Specialty Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Amal Jubran, Principal Investigator-Staff Physician, RML Specialty Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXJ014; R01NR016055 (NIH)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Muscle Weakness
Keywords: muscle strength; muscle function; functional status
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuro-muscular electrical stimulation (Active Comparator): Intervention:Neuromuscular electrical stimulation (NMES)
  NMES stimulation will be applied to lower extremity muscle groups up to 5 days a week until discharge. Standard physical therapy will also be administered by a therapist distinct from the therapist administering NMES
  Interventions: Device: Neuromuscular electrical Stimulation (NMES)
- Sham stimulation (Sham Comparator): Intervention: sham stimulation
  Sham stimulation will be applied to lower extremity muscle groups up to 5 days a week until discharge. Standard physical therapy will also be administered by a therapist distinct from the therapist administering sham-NMES
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Neuromuscular electrical Stimulation (NMES) — Electrical stimulation of lower extremities will be applied using an electrotherapy stimulator device (Vectra® Neo). The intensity of stimulation will be titrated based on maximal tolerable muscle contraction
  Arms: Neuro-muscular electrical stimulation
Device: Sham Stimulation — Sham stimulation of lower extremities will be applied using an electrotherapy stimulator device (Vectra® Neo).
  Arms: Sham stimulation

SUMMARY:
The primary aim of this proposal is to test the effectiveness of neuromuscular electrical stimulation (NMES) in improving functional status and muscle function in patients receiving prolonged mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Duration of mechanical ventilation >14 days
* Sufficiently awake
* Able to speak and comprehend English
* Willingness to participate

Exclusion Criteria:

* Cardiopulmonary Instability
* Acute-onset neuromuscular disease
* Lower-extremity amputee or paresis
* Open wound at electrode application points
* Pitting edema grade ≥3
* Presence of pacemaker, implanted defibrillator, or ventricular-assist device
* inability to transfer from sitting to standing before critical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Time to reach independence in performing functional activity | Hospital discharge, an expected average stay of 5 weeks
  Functional activity as measured by functional activity measurement for the ICU (FSS-ICU)

SECONDARY OUTCOMES:
The percentage of patients who can perform functional activities independently | Hospital discharge, an expected average stay of 5 weeks
  Percentage of patients with an FSS-ICU score ≥ 25 at discharge from LTACH

CONTACTS AND LOCATIONS:
Overall Officials: Amal Jubran, MD, Principal Investigator — RML Specialty Hospital
Locations (1):
- RML Specialty Hospital, Hinsdale, Illinois, United States

IPD SHARING:
Plan to Share IPD: No